CLINICAL TRIAL: NCT03723902
Title: Strength Training and Protein Supplementation in Pre-frail Elderly Individuals. Effects on Muscle Mass, Muscle Strength, Rate of Force Development and Functional Capacity
Brief Title: The Effect of Strength Training and Protein Supplementation in Old Pre-frail Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ST-PF
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Aging
Keywords: Strength training; Pre-frail
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training + protein supplement (Experimental): Heavy-load strength training, Protein supplementation
  Interventions: Other: Heavy-load strength training; Dietary Supplement: Protein supplementation
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Heavy-load strength training — Three weekly sessions of heavy-load strength training for 10 weeks
  Other Names: Resistance exercise
  Arms: Strength training + protein supplement
Dietary Supplement: Protein supplementation — Daily supplementation of 2 x 17 grams of milk protein
  Arms: Strength training + protein supplement

SUMMARY:
The aim of this study is to investigate the effects of a lower-body strength training regime combined with protein supplementation in pre-frail elderly individuals. Participants are randomized to a group performing three weekly sessions of heavy-load strength training for 10 weeks and receiving daily protein supplementation, or a non-training, non-supplemented control group. The endpoints are changes in body composition, the relative changes in different compartments of the quadriceps femoris muscles, and the relationships between changes in muscle mass, muscle thickness, strength, and functional capacity. The investigators hypothesize that 10 weeks of heavy load strength training and protein supplementation will elicit improvements in muscle mass, strength, and functional performance. Moreover, it is hypothesized that improvements in strength will correlate with the improvements in functional performance.

DETAILED DESCRIPTION:
Aging is accompanied by a loss of muscle mass and strength. Because muscle strength is associated with functional performance in elderly individuals, various tasks of daily living is hampered by the overall decline. The consequence is a vicious circle, where inactivity caused by reduced functional capacity accelerates the loss of muscle mass, strength and physical function. The Short Physical Performance Battery (SPPB) is commonly used to assess functional capacity, where individuals with a score of 10 or less out of maximum 12 may be categorized as pre-frail. Because small-to-moderate limitations in functional status assessed by SPPB is associated with higher odds of losing future mobility, these individuals represent a group of great interest. Strategies to improve functional capacity in this population are therefore important. It is established that heavy-load strength training, alone or in combination with protein supplementation, can improve muscle mass, strength, and function in elderly individuals. However, most studies have focused on healthy older adults, and less is known about the effects of heavy-load strength training in pre-frail elderly individuals. Moreover, the extent to which training-induced gains in muscle mass and size are related to improvements in strength and functional capacity is still poorly understood, because few intervention studies in this population have quantified hypertrophy precisely. Hence, the aim of this study is to investigate the effects of 10 weeks of heavy load strength training, performed three times per week, on muscle mass (DXA scan), muscle thickness (ultrasound), muscle strength (dynamic and isometric), rate of force development, chair rise ability, and gait velocity. Participants are randomized to a group performing three weekly sessions of heavy-load strength training or a control group. In addition, to optimize gains in muscle mass and strength, the strength training group will receive daily protein supplementation throughout the intervention period. The investigators hypothesize that the intervention will improve muscle mass, muscle thickness and strength, and that improvements in muscle strength and rate of force development will be correlated with improvements in functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 75
* Short Physical Performance Battery (SPPB) score ≤ 10

Exclusion Criteria:

* Lactose intolerance
* Milk allergy
* Diseases or musculoskeletal disorders contraindicating training/testing

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2015-12-21 (Actual)

PRIMARY OUTCOMES:
Muscle strength of m. Quadriceps Femoris | Change from baseline at 10 weks
  Maximal isometric muscle strength of m. quadriceps femoris (maximal voluntary contraction for the knee extensors)
Muscle strength of m. quadriceps femoris | Change from baseline at 10 weeks
  Maximal dynamic muscle strength of m. quadriceps femoris (knee extension 1 repetition maximum)
Leg lean mass | Change from baseline at 10 weeks
  Measured by Dual-energy X-ray Absorptiometry (DXA-scan)

SECONDARY OUTCOMES:
Total lean mass | Change from baseline at 10 weeks
  Measured by Dual-energy X-ray Absorptiometry (DXA-scan)
Fat mass | Change from baseline at 10 weeks
  Measured by Dual-energy X-ray Absorptiometry (DXA-scan)
Bone mineral density | Change from baseline at 10 weeks
  Measured by Dual-energy X-ray Absorptiometry (DXA-scan)
m. Vastus Lateralis thickness | Change from baseline at 10 weeks
  Measured by ultrasound
m. Rectus Femoris thickness | Change from baseline at 10 weeks
  Measured by ultrasound
m. Vastus Intermedius thickness | Change from baseline at 10 weeks
  Measured by ultrasound
m. Vastus Medialis thickness | Change from baseline at 10 weeks
  Measured by ultrasound
Isometric knee extension rate of force development (RFD max) | Change from baseline at 10 weeks
  Measured during maximal voluntary contraction
Isometric knee extension force at 100 ms | Change from baseline at 10 weeks
  Force at 100 ms during maximal voluntary contraction
Habitual gait velocity | Change from baseline at 10 weeks
  Time (sec) to walk 6 meters at preferred gait speed
Five times chair-rise performance | Change from baseline at 10 weeks
  Time (sec) to rise from a chair five times
Stair climbing | Change from baseline at 10 weeks
  Time (sec) to climb a staircase
Diet assessment | Change from baseline at 10 weeks
  24-hour diet recall interviews

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, Prof., Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No